CLINICAL TRIAL: NCT00355342
Title: A Randomized, Double-Blind, Parallel-Group Clinical Trial Evaluating the Effect of the Fluticasone Propionate/Salmeterol Combination Product 250/50mcg Twice Daily Via DISKUS® Inhaler Versus Salmeterol 50mcg Twice Daily Via DISKUS® Inhaler on Bone Mineral Density in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Bone Mineral Density Study In Patients With Chronic Obstructive Pulmonary Disease. DISKUS® Inhaler is a Trademark of the GSK Group of Companies.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCO40041
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Osteoporosis; Bone Mineral Density; Osteopenia; Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Osteoporosis; Bone Diseases, Metabolic | interventions — Salmeterol Xinafoate; BID protein, human; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Salmeterol 50 mcg BID (Experimental): Participants randomized to this arm received salmeterol 50 microgram (mcg), formulated with lactose via the DISKUS™ inhaler one inhalation twice daily (BID) one inhalation in the morning and one inhalation in the evening for 156 Weeks. Each DISKUS contained 60 doses of study medication. Participant were provided with albuterol/salbutamol as relief medication. DISCUS is registered trademark product of GlaxoSmithKline.
  Interventions: Drug: Salmeterol 50 mcg BID; Device: DISKUS inhaler
- Fluticasone Propionate/Salmeterol 250/50 mcg BID (Experimental): Participants randomized to this arm received Fluticasone propionate/salmeterol combination product 250/50 mcg, formulated with lactose via the DISKUS inhaler one inhalation BID, one inhalation in the morning and one inhalation in the evening for 156 Weeks. Each DISKUS contained 60 doses of study medication. Participant were provided with albuterol/salbutamol as relief medication.
  Interventions: Drug: Fluticasone Propionate/Salmeterol 250/50 mcg BID; Device: DISKUS inhaler

INTERVENTIONS:
Drug: Salmeterol 50 mcg BID — Salmeterol xinafoate 50 mcg strength DISKUS inhaler (formulated with lactose), BID in the morning and evening.
  Other Names: GR33343G
  Arms: Salmeterol 50 mcg BID
Drug: Fluticasone Propionate/Salmeterol 250/50 mcg BID — Fluticasone propionate/salmeterol xinafoate combination product 250/50mcg strength DISKUS inhaler (formulated with lactose), BID in the morning and evening.
  Other Names: CCI18781/GR33343G
  Arms: Fluticasone Propionate/Salmeterol 250/50 mcg BID
Device: DISKUS inhaler — Each participant received study medication via the DISKUS, for one of two possible treatment groups. Each DISKUS contained 60 doses of study medication. Participants were instructed to administer medication BID (one inhalation in the morning and one inhalation in the evening) approximately 12 hours apart for 156-week treatment period.

SUMMARY:
This study will last up to 3 years. You will visit the clinic up to 14 times. Certain visits will include lung function tests and scans of your bones. The purpose of this study is to determine the effect of the steroid component of an inhaled product on bone mineral density in patients with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion criteria:

* Established clinical history of COPD.
* Baseline FEV1 <70% predicted normal, and FEV1/FVC ratio of less than 70%.
* Smoking history of at least 10 pack-years, where both current and former smokers will be eligible.
* Must have at least one native, evaluable hip.

Exclusion criteria:

* History of or evidence for metabolic bone diseases other than osteoporosis or osteopenia.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2004-04-28 (Actual); Primary Completion 2007-09-06 (Actual); Study Completion 2007-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- United States (34):
  - GSK Investigational Site, Berkeley, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, North Chicago, Illinois
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Cadillac, Michigan
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Bronxville, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Milan, Tennessee
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: SCO40041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SCO40041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCO40041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SCO40041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SCO40041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SCO40041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SCO40041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 186 participants, with chronic obstructive pulmonary disease (COPD) were randomized at 31 centers in the United States. Study duration was 14-21 day Single-Blind Run-In period, 156-week treatment period and follow-up phone contact within 2 weeks of treatment stop.
Pre-assignment Details: A total of 247 participants were screened for this study, of whom 61 were screen failures and 186 participants were randomized in the study.
Period: Overall Study
Arm/Group | Salmeterol 50 mcg BID | Fluticasone Propionate/Salmeterol 250/50 mcg BID
Started | 94 | 92
Completed | 55 | 56
Not Completed | 39 | 36
Not completed — Adverse Event | 13 | 15
Not completed — Lost to Follow-up | 4 | 2
Not completed — Withdrawal by Subject | 14 | 11
Not completed — Sponsor terminated study | 2 | 2
Not completed — Overcompliant-PI discretion | 1 | 0
Not completed — Use of prohibited medication | 1 | 0
Not completed — COPD exacerbation | 1 | 1
Not completed — Dispensed wrong study drug kit | 1 | 0
Not completed — Non-compliance with Dexa scans | 1 | 0
Not completed — Withdrawal by participant and physician | 1 | 0
Not completed — Participant relocated | 0 | 1
Not completed — Participant discontinued study drug | 0 | 1
Not completed — Study management | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Use of protocol excluded medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Salmeterol 50 mcg BID: Participants randomized to this arm received salmeterol 50 mcg, formulated with lactose via the DISKUS inhaler one inhalation BID one inhalation in the morning and one inhalation in the evening for 156 Weeks. Each DISKUS contained 60 doses of study medication. Participant were provided with albuterol/salbutamol as relief medication.
- Total: Total of all reporting groups
Arm/Group | Salmeterol 50 mcg BID | Fluticasone Propionate/Salmeterol 250/50 mcg BID | Total
Number analyzed (Participants) | 94 | 92 | 186
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (9.52) | 65.4 (8.36) | 65.6 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 59 | 55 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Hispanic | 1 | 0 | 1
  Race: Black | 1 | 4 | 5
  Race: South Asian | 0 | 1 | 1
  Race: White/Caucasian | 92 | 87 | 179

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) at the Lumbar Spine L1-L4
Description: BMD, a measure of bone density, reflecting the strength of bones as represented by calcium content. The BMD test detects osteopenia (mild bone loss) and osteoporosis (more severe bone loss, which may cause symptoms). BMD at the lumber spine (L1-L4) was measured via dual energy x-ray absorptiometry (DEXA) (using DEXA equipment) scans at Baseline and every 26 weeks during the study. Acceptable DEXA measurements must be conducted prior to the first dose of randomized study medication. Baseline was defined as the collections taken on Day 1 of treatment period. Change from Baseline was calculated by subtracting the Baseline value from indicated time point value.
Time Frame: Baseline and Week 26, 52, 78, 104, 130, and 156
Population: The Safety population - Safety population was defined as all randomized participants who are at least 50% compliant with taking study drug and have a post-Baseline BMD scan. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Salmeterol 50 mcg BID | Fluticasone Propionate/Salmeterol 250/50 mcg BID
Number analyzed (Participants) | 84 | 82
Percent Change
  Week 26: number analyzed (Participants) | 79 | 80
  Week 26 | 0.5 (0.33) | 0.2 (0.40)
  Week 52: number analyzed (Participants) | 68 | 68
  Week 52 | 0.8 (0.39) | 1.3 (0.43)
  Week 78: number analyzed (Participants) | 57 | 64
  Week 78 | 1.3 (0.52) | 1.0 (0.64)
  Week 104: number analyzed (Participants) | 54 | 62
  Week 104 | 0.9 (0.55) | 0.8 (0.71)
  Week 130: number analyzed (Participants) | 53 | 58
  Week 130 | 0.3 (0.66) | 1.0 (0.81)
  Week 156: number analyzed (Participants) | 51 | 57
  Week 156 | 0.3 (0.68) | 1.9 (0.88)
Statistical Analysis 1: Comparison: Salmeterol 50 mcg BID vs Fluticasone Propionate/Salmeterol 250/50 mcg BID; The analysis is presented for slope estimate calculated for the percent change from Baseline values at Week 26, 52, 78, 104, 130, and 156; Test type: Equivalence — The null hypothesis for the primary measure is that the difference between the effects of fluticasone propionate/salmeterol combination product 250/50mcg BID and salmeterol 50mcg BID on the change in BMD assessed at the L1-L4 region of the spine is greater than 1 %/year; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [0.06 to 1.49], Standard Error of Mean 0.36 — Analysis Model: Percent change from baseline BMD = treatment + time (years) + treatment*time + baseline BMD + sex + investigator + age + BMI + FEV1 severity + b/l activity level + b/l calcium supp. use + smoking status; Age split by category (40-64 years old, 65 or older). FEV1 severity based on GOLD Stage (Mild/Moderate, Severe/Very Severe). Activity based on 0-10 Physical Activity Scale (split by median, <7, >=7). Slope estimates based on treatment*time via repeated measures model with unstructured covariance

2. Secondary Outcome: Percent Change From Baseline in BMD at the Total Hip
Description: BMD, a measure of bone density, reflecting the strength of bones as represented by calcium content. The BMD test detects osteopenia (mild bone loss) and osteoporosis (more severe bone loss, which may cause symptoms).BMD at the total hip was measured via dual energy x-ray absorptiometry (DEXA) (using DEXA equipment) scans at Baseline and every 26 weeks during the study. Acceptable DEXA measurements must be conducted prior to the first dose of randomized study medication. Baseline was defined as the collections taken on day 1 of treatment period. Change from Baseline was calculated by subtracting the Baseline value from indicated time point value.
Time Frame: Baseline and Week 26, 52, 78, 104, 130, and 156
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Salmeterol 50 mcg BID | Fluticasone Propionate/Salmeterol 250/50 mcg BID
Number analyzed (Participants) | 84 | 82
Percent Change
  Week 26: number analyzed (Participants) | 78 | 80
  Week 26 | -0.3 (0.28) | -0.4 (0.31)
  Week 52: number analyzed (Participants) | 67 | 69
  Week 52 | -0.5 (0.32) | -1.4 (0.35)
  Week 78: number analyzed (Participants) | 56 | 64
  Week 78 | -0.8 (0.45) | -2.1 (0.46)
  Week 104: number analyzed (Participants) | 55 | 62
  Week 104 | -1.1 (0.46) | -2.6 (0.50)
  Week 130: number analyzed (Participants) | 53 | 58
  Week 130 | -1.7 (0.47) | -2.7 (0.44)
  Week 156: number analyzed (Participants) | 51 | 57
  Week 156 | -1.8 (0.57) | -2.9 (0.46)
Statistical Analysis 1: Comparison: Salmeterol 50 mcg BID vs Fluticasone Propionate/Salmeterol 250/50 mcg BID; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.78 to 0.24], Standard Error of Mean 0.26 — [estimate comment as in outcome 1, analysis 1]; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 160 weeks
Description: Intent-to-treat population was defined as all randomized participants receiving at least one dose of study drug and was analyzed according to the treatment each participant was scheduled to have received.
Arm/Group | Salmeterol 50 mcg BID | Fluticasone Propionate/Salmeterol 250/50 mcg BID
All-Cause Mortality (participants affected / at risk) | 7/94 | 5/92
Serious Adverse Events (participants affected / at risk) | 33/94 | 32/92
Other Adverse Events (participants affected / at risk) | 63/94 | 72/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Salmeterol 50 mcg BID (N=94) | Fluticasone Propionate/Salmeterol 250/50 mcg BID (N=92)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 | 11
Pneumonia (Infections and infestations) | 4 | 6
Myocardial infarction (Cardiac disorders) | 0 | 5
Chest pain (General disorders) | 1 | 2
Coronary artery disease (Cardiac disorders) | 3 | 0
Lobar pneumonia (Infections and infestations) | 2 | 1
Syncope (Nervous system disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Diverticulitis (Infections and infestations) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Asthenia (General disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cor pulmonale (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pain (General disorders) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Renal artery occlusion (Renal and urinary disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Ulcer haemorrhage (General disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Whiplash injury (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salmeterol 50 mcg BID (N=94) | Fluticasone Propionate/Salmeterol 250/50 mcg BID (N=92)
Nasopharyngitis (Infections and infestations) | 21 (38) | 28 (48)
Sinusitis (Infections and infestations) | 15 (23) | 12 (22)
Upper respiratory tract infection (Infections and infestations) | 11 (13) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 8 (9)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 10 (14)
Bronchitis (Infections and infestations) | 7 (7) | 8 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (10)
Headache (Nervous system disorders) | 6 (6) | 8 (11)
Hypertension (Vascular disorders) | 6 (6) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 4 (5)
Influenza (Infections and infestations) | 4 (4) | 6 (7)
Anxiety (Psychiatric disorders) | 4 (4) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Oral candidiasis (Infections and infestations) | 4 (6) | 5 (11)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (7)
Candidiasis (Infections and infestations) | 1 (1) | 7 (12)
Fatigue (General disorders) | 3 (3) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (6)
Oedema peripheral (General disorders) | 6 (9) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 5 (5)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 5 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7)
Pain (General disorders) | 5 (5) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.